CLINICAL TRIAL: NCT05627609
Title: Sunlight-mediated Inter-organ Leukocyte Exchange
Acronym: SMILE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Responsible Party: Principal Investigator, Nicholas Schwab, Prof. Dr. rer. nat., University Hospital Muenster
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SMILE-2022-439-f-S
Record Dates: First submitted 2022-11-16; First posted 2022-11-25 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Multiple Sclerosis
Keywords: UVB; scRNAseq
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants with high Vitamin D genotype risk score (Experimental)
  Interventions: Device: 311 nm narrowband UVB irradiation
- PArticipants with low Vitamin D genotype risk score (Experimental)
  Interventions: Device: 311 nm narrowband UVB irradiation

INTERVENTIONS:
Device: 311 nm narrowband UVB irradiation — Participants will be irradiated with 311nm UVB for 5 days per week and 4 weeks in total.

SUMMARY:
Ultraviolet B (UVB) irradiation induces regulatory immune cell types that may transmigrate from the skin to the blood and to the central nervous system and exert regulatory effects. Vitamin D deficiency-associated gene variants should reduce this effect if this is mediated by vitamin D. For this study, participants will be irradiated with UVB for 4 weeks. Single cell RNA Sequencing will be performed on isolated immune cells from skin, blood and Cerebrospinal fluid (CSF), before and after irradiation.

DETAILED DESCRIPTION:
The aim of this study will be to increase the Vitamin D3-serum concentrations in Multiple Sclerosis patients via UVB radiation with regard to different Vitamin D deficit-associated genotypes and analyse the effects of Vitamin D increase and UVB radiation, in general, on their immune cells. Participants of this study will be recruited from the pool of already registered MS patients at the department of neurology at the UKM and from resident practitioners of the Neuroimmunologisches Kompetenznetzwerk Münsterland. The UVB radiation of the participants will take place during wintertime to avoid any interference by ambient sunlight. As the participants will not take any supplements of Vitamin D, their serum concentration should be very low. The participants will be screened beforehand for their Vitamin D deficit-associated single nucleotide polymorphism and sorted into two groups depending on their calculated risk scores. The patients will also receive a clinical assessment in the department of neurology and dermatology and a cranial MRT. 17 patients each will be sorted into one of two groups: either Vitamin D deficiency high-risk or low-risk. The UVB influence on Vitamin D-serum concentration increases between those two groups should then be dependent on the associated genotypes. We will track those changes by taking blood samples before and after the radiation. We will also take samples of the skin and, for participants opting in, cerebrospinal fluid (CSF). This will allow us to isolate single cells from each of the three compartments and sequence them on a RNA transcriptomic level following the 10x workflow. UVB radiation will induce immunomodulating effects in the skin and Vitamin D was shown to be one of those effects, as its synthesis is initiated by UVB radiation and its binding to Vitamin D receptors renders immune cells more regulatory. If differences in immune cell alterations were found between the two groups of risk scores, they should be attributed to the associated genotypes, shedding new light on the influence of Vitamin D on the pathogenesis of MS patients and on the immune system in general.

By utilizing single-cell RNA-sequencing on isolated immune cells of those three compartments, before and after the UVB radiation, we will be able to have a relatively unbiased approach to investigating the influence of UVB radiation and, separately, Vitamin D on the immune cells. Specific cell signatures of sequenced immune cells from the three compartments will allow us to track the migration of the induced cells from the skin through the blood and into the CSF. Additionally, CSF and serum isolated from blood will be assessed for Epstein-Barr-Virus antibody titers and extracellular vesicles. All this data will contribute to our multidimensional analysis using bioinformatics workflows based on linear methods such as principal components analysis and non-linear tools based on neural networks and Bayesian variational inference.

ELIGIBILITY:
Inclusion Criteria:

* RRMS according to revised McDonald criteria (2017) or healthy volunteer
* Patients under treatment of natalizumab, teriflunomide, glatirameracetat or dimethyl fumarate for at least 4 weeks of therapy, or therapy-naïve patients will be included

Exclusion Criteria:

* Patients receiving treatment in the last 3 months of interferon-β, fingolimod, alemtuzumab, ocrelizumab, cladribine, ofatumumab, ozanimod, or ponesimod
* Vitamin D supplementation in the last 8 weeks
* UVB-narrowband contraindicated skin diseases (e.g., cutaneous neoplasia)
* Lacking the ability to stand on their own in the treatment chamber
* Signs of intolerance regarding UVB radiation
* Intake of UV-sensitive therapeutics
* Further autoimmune diseases (e.g., Morbus Crohn, psoriasis, neurodermatitis)
* Additional recreational or therapeutic UV radiation (e.g., solarium)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Vitamin D3 serum concentration (ng/mL) | 4 weeks
  Changes in Vitamin D3 serum concentration (ng/mL) of RRMS patients with regard to different Vitamin D3 deficit-associated genotypes before and after UVB-narrowband radiation.

SECONDARY OUTCOMES:
single-cell RNA sequencing | 1 year
  By utilizing single-cell RNA sequencing of immune cells from the skin and blood and even potentially the cerebrospinal fluid (CSF) we want to analyze the phenotype of UVB-induced immune cells and potentially track their migration from the skin through the peripheral blood into the CSF. If any of the witnessed immune regulatory effects in those three compartments can be attributed to the increase of Vitamin D3 through UVB radiation, we should be able to differentiate those effects among the different genotypes. Since MS risk and severity correlate with EBV infection and infectious mononucleosis, we will also measure EBV antibody titers before and after UVB radiation in blood and CSF.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Muenster, Münster, North Rhine-Westphalia, Germany